CLINICAL TRIAL: NCT02410668
Title: The Effects of Flaxseed Supplement on Weight, Lipid Profile and Inflammatory Factors in Overweight and Obese Subjects
Brief Title: The Effects of Flaxseed Supplement on Weight and Biochemical Factors in Overweight and Obese Subject
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flaxseed (Active Comparator): 30 grams Flaxseed powder combine with dietary and exercise recommendation
  Interventions: Dietary Supplement: flaxseed; Behavioral: Exercise recommendation
- control (Placebo Comparator): dietary and exercise recommendation
  Interventions: Dietary Supplement: Placebo; Behavioral: Exercise recommendation

INTERVENTIONS:
Dietary Supplement: flaxseed
  Arms: Flaxseed
Dietary Supplement: Placebo
  Arms: control
Behavioral: Exercise recommendation

SUMMARY:
To study the effects of Flaxseed supplement on weight, lipid profile and inflammatory factors in subjects with over weight and obesity, 50 patients will be randomly allocated to receive placebo or 30 grams milled Flaxseed for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, weight, waist and hip circumference, lipid profile and some inflammatory markers will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40

Exclusion Criteria:

* diabetes mellitus
* cardiovascular diseases and cancers
* major systemic diseases
* gastrointestinal problems
* liver and renal failure
* history of allergy or high consumption of nuts, flaxseed, or sesame seeds
* weight loss within the past 6 mo of >5% of body weight or current adherence to a weight-reduction diet
* pregnancy, lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
weight | 12 weeks
waist and hip circumference | 12 weeks

SECONDARY OUTCOMES:
lipid profile | 12 weeks

REFERENCES:
- [Derived] Yari Z, Rahimlou M, Poustchi H, Hekmatdoost A. Flaxseed supplementation improves anthropometric measurements, metabolic, and inflammatory biomarkers in overweight and obese adults. Int J Vitam Nutr Res. 2022 Jul;92(3-4):161-168. doi: 10.1024/0300-9831/a000565. Epub 2019 Mar 7. PMID 30843767